CLINICAL TRIAL: NCT04831489
Title: Risk of Pulmonary Micro-aspiration in Intubated vs Sedated Patients Undergoing ERCP
Brief Title: Microaspiration in ERCP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Moshira sayed mohamed, Lecturer of Anasthesia and intensive care, Theodor Bilharz Research Institute
Other Study IDs: Microaspiration in ERCP
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Pulmonary Microaspiration
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- deep sedation: Anesthesia will be induced using titrated doses of propofol (0.5-1.5 mg/kg) and fentanyl (25-50 μg) initially to carefully maintain spontaneous breathing yet maintaining airway patency. Once adequate jaw relaxation is achieved, the endoscopy probe will be inserted. Maintenance of sedation will be carried out using propofol infusion between 80-120 mcg/kg/min. Additional dose 25-50 mg propofol will be given to the patient if spontaneous movement occurs
  Interventions: Radiation: Imaging
- Genral anesthesia: After mask pre-oxygenation, anesthesia will be induced with (2 mg/kg) propofol and (1 μg /kg) fentanyl. The neuromuscular blockade will be achieved with (0.5 mg/kg) atracurium followed by tracheal intubation. Anesthesia will be maintained to keep the end-tidal anesthetic concentrations within 1 MAC for sevoflurane.
  The neuromuscular blockade will be maintained with intermittent doses of atracurium (0.1mg/kg). Mechanical ventilation is adjusted with fresh gas flow oxygen in air 30-40% at a rate of 2 L/min to maintain end-tidal carbon dioxide of 35-40 mm Hg. Reversal of neuromuscular blockade will be achieved by intravenous administration of neostigmine 0.05 mg/kg and atropine 0.02 mg/kg.
  Interventions: Radiation: Imaging

INTERVENTIONS:
Radiation: Imaging — pre and postoperative CT scan of lung

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) is considered the gold standard in diagnosing and treating biliary and pancreatic diseases. Patients planned for ERCP often have additional comorbidities that make them high-risk candidates for general anesthesia so; the optimized choice of the anesthetic technique represents a real challenge. apparent aspiration is noticeable however microaspiration is hard to detect clinically. our study aims at determining whether general anesthesia with endotracheal intubation or deep sedation is safer in ERCP patients.

DETAILED DESCRIPTION:
Endoscopic retrograde cholangiopancreatography (ERCP) is considered the gold standard in diagnosing and treating biliary and pancreatic diseases. In fact, with the wide use of ERCP, many critical patients in whom conventional surgery was a high-risk procedure could be managed by endoscopic treatment.

Compared to other endoscopic procedures, ERCP is considered a relatively longer and more complex one, with a substantially higher complication rate. Anesthetic techniques must facilitate the success of this procedure without adding to morbidity.

Patients planned for ERCP often have additional comorbidities that make them high-risk candidates for general anesthesia so; the optimized choice of the anesthetic technique represents a real challenge.

Many anesthetic techniques are used, ranging from conscious sedation to general anesthesia. The worldwide accepted method is deep sedation in the presence of an anesthetist without endotracheal intubation. Intubation is recommended in very exceptional cases, for example is morbidly obese patients.

According to some authors, general anesthesia is less used as an anesthetic technique in ERCP; drawbacks of GA include: the lengthier time required for induction of and recovery from anesthesia which affects patients' turnover, the risk of residual neuromuscular blockade, the higher cost as well as ERCP is usually a day case procedure favoring the sedation technique. On the other hand, monitored anesthesia care or deep sedation in remote locations can avoid these drawbacks.

For ERCP cases, which can be very challenging, few studies have addressed what is the best anesthetic choice, i.e. deep sedation or general anesthesia with intubation. Significant complications such as aspiration, hypoxemia, and hypotension are potential risks in patients undergoing ERCP procedures, and important factors that can modify these events' severity include patients' ASA status, patients' hydration and oxygenation status, and monitoring techniques used during the procedure.

Perioperative pulmonary aspiration (POPA) may lead to clinically significant morbidities and/or mortality. The risk factors for pulmonary aspiration are usually overlooked unless the patient has a history of gastrointestinal diseases (for example gastroesophageal reflux disease, upper gastrointestinal bleeding, or intestinal obstruction). However, aspiration pneumonia is seldom observed in healthy patients undergoing regular endoscopy. On the other hand, prolonged or difficult procedures may be associated with increased risks of regurgitation and aspiration.

Apparent aspiration is a notable adverse event during gastrointestinal endoscopy, on the other hand, microaspiration is an underreported complication, and data about it is scarce. Since hypoxemia is a common manifestation of pulmonary aspiration and pulse oximetry monitoring is a routine practice, therefore, postoperative hypoxemia (POH) can be used as a potential signal for POPA.

There is no conclusive data to support or refuse the need for endotracheal intubation to avoid microaspiration during ERCP; therefore, the participants in the study decided to prospectively compare both techniques as regards the risk of microaspiration.

ELIGIBILITY:
Inclusion Criteria:

1. ASA 1-3.
2. Age above 18 years old.
3. Preoperative pulmonary stability criteria (defined as a respiratory rate 12-24 breaths per minute, SpO2 ≥ 94% on room air) -

Exclusion Criteria:

1. Age < 18 years.
2. Morbid obesity BMI ≥ 40 Kg/ m2.
3. Pregnancy.
4. Fasting ≤ 6 hours for solid food and ≤ 2 hours for clear liquids. 4
5. A pre-existing lung condition in patients requiring supplemental oxygen, inhalational bronchodilator, or systemic bronchodilator or steroid.
6. Patients in the intensive care unit and/or requiring mechanical ventilation prior to the procedure.
7. Previously intubated patients during the same hospitalization.
8. Tracheostomized patients.
9. Patients with swallowing disorders.
10. Bowel obstruction.
11. Anticipated difficult intubation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the population of the study will be randomly selected from the daily scheduled cases undergoing ERCP in the Gastroenterology department of Theodor Bilhrarz research institute.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
POPA | 24 hours postoperatively
  Perioperative Pulmonary Aspiration (POPA), which will be defined as the presence of an acute pulmonary infiltrate on chest CT within the 24 hours period following ERCP.

SECONDARY OUTCOMES:
Number of intraoperative hypoxic episodes. | 24 hours postoperative.
  Number of intraoperative hypoxic episodes in postoperative period

CONTACTS AND LOCATIONS:
Locations (1):
- Theodor Bilharz research institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shah SK, Mutignani M, Costamagna G. Therapeutic biliary endoscopy. Endoscopy. 2002 Jan;34(1):43-53. doi: 10.1055/s-2002-19395. PMID 11778129
- [Background] Motiaa Y, Bensghir M, Jaafari A, Meziane M, Ahtil R, Kamili ND. Anesthesia for endoscopic retrograde cholangiopancreatography: target-controlled infusion versus standard volatile anesthesia. Ann Gastroenterol. 2016 Oct-Dec;29(4):530-535. doi: 10.20524/aog.2016.0071. Epub 2016 Jul 14. PMID 27708522
- [Background] Garewal D, Vele L, Waikar P. Anaesthetic considerations for endoscopic retrograde cholangio-pancreatography procedures. Curr Opin Anaesthesiol. 2013 Aug;26(4):475-80. doi: 10.1097/ACO.0b013e3283620139. PMID 23635608
- [Background] Mazanikov M, Udd M, Kylanpaa L, Lindstrom O, Aho P, Halttunen J, Farkkila M, Poyhia R. Patient-controlled sedation with propofol and remifentanil for ERCP: a randomized, controlled study. Gastrointest Endosc. 2011 Feb;73(2):260-6. doi: 10.1016/j.gie.2010.10.005. PMID 21295639
- [Background] Sorser SA, Fan DS, Tommolino EE, Gamara RM, Cox K, Chortkoff B, Adler DG. Complications of ERCP in patients undergoing general anesthesia versus MAC. Dig Dis Sci. 2014 Mar;59(3):696-7. doi: 10.1007/s10620-013-2932-2. Epub 2013 Nov 8. No abstract available. PMID 24202650
- [Background] Barnett SR, Berzin T, Sanaka S, Pleskow D, Sawhney M, Chuttani R. Deep sedation without intubation for ERCP is appropriate in healthier, non-obese patients. Dig Dis Sci. 2013 Nov;58(11):3287-92. doi: 10.1007/s10620-013-2783-x. Epub 2013 Jul 23. PMID 23877477